CLINICAL TRIAL: NCT03003949
Title: The Menopause Transition: Estrogen Variability, HPA Axis and Affective Symptoms
Brief Title: The Menopause Transition: Estrogen Variability, Stress Reactivity and Mood
Acronym: Changes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: In-person visit restrictions due to COVID-19
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-1731; 1R01MH108690-01A1 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-28 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2020-03

CONDITIONS: Perimenopausal Disorder; Stress, Emotional
Keywords: perimenopause; menopause transition; estrogen; stress; mood
MeSH Terms: conditions — Stress, Psychological | interventions — Estradiol; Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Patch and Placebo Capsule (Placebo Comparator): Placebo patches worn for 16 weeks. On the 9th week of patch, oral placebo capsule taken daily for 12 days. Following the 16 weeks of patch use oral placebo capsule taken daily for 12 days.
  Interventions: Drug: Placebo Patch; Drug: Placebo Oral Capsule
- Estradiol patch and progesterone capsule (Active Comparator): Estradiol patches worn for 16 weeks. On the 9th week of patch, oral progesterone capsule taken daily for 12 days. Following the 16 weeks of estradiol patch use oral progesterone capsule taken daily for 12 days.
  Interventions: Drug: Estradiol Patch, 0.1 Mg/24 Hours Weekly Transdermal Film, Extended Release; Drug: Progesterone Capsule

INTERVENTIONS:
Drug: Estradiol Patch, 0.1 Mg/24 Hours Weekly Transdermal Film, Extended Release — Transdermal Estradiol worn daily for 16 weeks (patch changed every 7 days).
  Other Names: Climara; Prometrium
  Arms: Estradiol patch and progesterone capsule
Drug: Placebo Patch — Matching placebo patches to be worn every day for 16 weeks (patch changed every 7 days).
  Other Names: Placebos
  Arms: Placebo Patch and Placebo Capsule
Drug: Progesterone Capsule — Micronized progesterone (200 mg) will be administered every day for 12 days during the 9th week of randomization and again following randomization at the 17th week
  Other Names: Progesterone
  Arms: Estradiol patch and progesterone capsule
Drug: Placebo Oral Capsule — Matching placebo capsules will be administered orally every day for 12 days during the 9th week of randomization and again following randomization at the 17th week.
  Other Names: Placebos
  Arms: Placebo Patch and Placebo Capsule

SUMMARY:
Women in the menopause transition ('perimenopause') are exposed to extreme hormone variability, tend to experience a unique set of severe stressors (e.g., divorce, death of loved ones), and are also at substantially elevated risk to suffer from mood and anxiety disorders. The purpose of this research is to understand the mechanisms by which variability in estradiol (E2) is associated with the symptoms of anxiety and anhedonia (loss of interest and pleasure - a common symptom of depression). By stabilizing E2 variability with a hormonal manipulation, this research will determine the degree to which the E2 variability (or E2 levels) plays a causal role in perimenopausal anxiety and anhedonia symptoms and whether it does so by affecting biological responses to stress.

DETAILED DESCRIPTION:
Framed within a diathesis-stress model, the primary objective of this research is to determine the pathophysiological mechanisms of estradiol (E2) in the clinical anxiety and anhedonia seen in the menopause transition (MT). Specifically whether E2 variability or E2 levels predict exaggerated hypothalamic-pituitary-adrenal (HPA) axis reactivity and impaired recovery to stress and, in turn, deficits in behavioral indices of threat responsivity and approach motivation and symptoms of anxiety and anhedonia. The secondary objective of the research is to use a hormonal manipulation as a mechanistic probe to stabilize E2 variability in premenopausal ranges and determine if: a) HPA axis reactivity/recovery represents a biomarker of behavioral and symptom responses to E2 stabilization; b) whether recent severe life stress predicts the HPA axis response to hormone stabilization.

A total of 170 women in the early or late MT who are eligible for the hormonal probe will be recruited to reflect the full continuum of anxiety and anhedonia symptoms based on self-report to the State-Trait Anxiety Inventory and the Snaith-Hamilton Pleasure Scale, respectively. However, the investigators will over-represent the clinically impairing end of the anxious and anhedonic phenotype (75% of the sample). Over an 8-week baseline, anxiety and anhedonia symptoms and serum E2 measured by liquid chromatography-tandem mass spectrometry (LC-MS/MS) will be assessed on a weekly basis. At baseline week 8, HPA axis (plasma cortisol and ACTH) response to the Trier Social Stress Test and behavioral measures of threat responsivity (via Dot-Probe task) and approach motivation (Effort Expenditure for Rewards Task 'EEfRT') will be determined. Using transdermal E2 as a pharmacological probe to stabilize variability of E2 in premenopausal ranges, women will then be randomized to transdermal E2 (0.10 mg) or placebo for 16 weeks. This is not a clinical efficacy trial. The investigators will use an randomized control trial (RCT) design with a hormonal manipulation in order to investigate the pathophysiologic role of E2 variability (or E2 levels) in HPA axis dysregulation and, in turn, threat responsivity and approach motivation. Serum E2 will be assessed weekly during weeks 9-16, and HPA axis reactivity to stress and behavioral responses to the Dot-Probe and EEfRT tasks will be assessed every four weeks during the 16 week probe.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal (either early perimenopause, defined as menstrual cycle length 7+ days longer or shorter than usual; or the late perimenopause, defined as ≥2 skipped cycles and an interval of amenorrhea ≥60 days but within one year of the last menstrual period)
* 45 to 60 years of age
* must be medically healthy

Exclusion Criteria:

* a history of cardiovascular disease (CVD) including coronary artery disease, arteriosclerosis, heart attack, or stroke
* Type I or II diabetes
* personal history of thrombotic events
* personal or family history suggesting elevated risk for E2-related cancer
* currently experiencing migraine headaches with aura

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Girdler, PhD, Principal Investigator — Research Professor
Locations (2):
- United States (2):
  - UNC SHARRP Lab, Chapel Hill, North Carolina
  - Susan Girdler, PhD, Principal Investigator, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit data to the Research Domain Criteria Database (RDoCdb) and/or the National Database for Clinical Trials Related to Mental Illness (NDCT). The investigators will work with RDoCdb and NDCT staff to define data structures for any data being collected as part of the study. Descriptive data will be submitted two times per year and provide supporting documentation as necessary for others to more fully understand the manner in which data were collected. The investigators will submit cumulative data each submission cycle and will review data for any personally identifiable information and ensure that data are loaded correctly. The investigators will share data within 4 months after submission and submit experimental data within 12 months after study completion. Study data for each publication will be created and submit a link to the RDoCdb study along with any publications so readers of articles can link back to the data used in RDoCdb and NDCT.

REFERENCES:
- [Derived] Lozza-Fiacco S, Gordon JL, Andersen EH, Kozik RG, Neely O, Schiller C, Munoz M, Rubinow DR, Girdler SS. Baseline anxiety-sensitivity to estradiol fluctuations predicts anxiety symptom response to transdermal estradiol treatment in perimenopausal women - A randomized clinical trial. Psychoneuroendocrinology. 2022 Sep;143:105851. doi: 10.1016/j.psyneuen.2022.105851. Epub 2022 Jul 2. PMID 35809362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Started | 40 | 42
Week 8 | 40 | 42
Week 16 | 38 | 35
Week 20 | 35 | 33
Week 24 | 35 | 32
Completed | 35 | 32
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.40 (2.52) | 49.39 (3.04) | 49.88 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 37 | 39 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 34 | 30 | 64
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in the Anxiety Score From State-Trait Anxiety Inventory
Description: The State-Trait anxiety inventory is consists of 20 questions on a 4-point force-choice Likert-type response scales (scores 0 - 3). The 20 questions are summed together for final score. The score can range from 0 to 60 with higher scores representing higher levels of anxiety. Change over time is defined as the difference in the least square means between timepoints and 95% confidence interval limits.
Time Frame: Baseline (Week 8), Weeks 16, 20 and 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Number analyzed (Participants) | 40 | 42
score on a scale
  Baseline (Week 8) to Week 16 | 2.74 [-4.08 to 9.57] | -0.89 [-6.47 to 4.67]
  Week 16 to Week 20 | -3.50 [-10.56 to 3.56] | 0.19 [-5.75 to 6.12]
  Week 20 to Week 24 | 3.63 [-3.57 to 10.83] | 3.75 [-2.24 to 9.73]

2. Primary Outcome: Change Over Time in Anhedonia Score From Snaith-Hamilton Pleasure Scale
Description: Anhedonia will be assessed using SHAPS scores which range from 14-56, with higher scores corresponding to higher levels of anhedonia. Change over time is defined as the difference in least square means between time points and 95% confidence interval limits.
Time Frame: Baseline (Week 8), Weeks 16, 20 and 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Number analyzed (Participants) | 40 | 42
score on a scale
  Baseline (Week 8) to Week 16 | -0.01 [-1.04 to 1.03] | -0.63 [-1.71 to 0.46]
  Week 16 to Week 20 | 0.12 [-0.87 to 1.27] | 0.88 [-0.27 to 2.03]
  Week 20 to Week 24 | 0.29 [-0.79 to 1.38] | -0.07 [-1.22 to 1.08]

3. Secondary Outcome: Change Over Time in AUC Cortisol Stress Response
Description: The stress biomarker cortisol (µg/dL) assessed at rest and in response to the Trier Social Stress test (AUC with respect to ground) at baseline (Week 8) and again post-randomization at weeks 16, 20 and 24. Blood serum samples for measuring cortisol are taken at immediately before the Trier Social Stress test and at 10, 20, 30, and 45 minutes post test. Change over time is defined as the difference in least square means between timepoints and with 95% confidence interval limits.
Time Frame: Baseline (Week 8), Weeks 16, 20 and 24
Population: Data reported for all samples collected.
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/dL
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Number analyzed (Participants) | 31 | 33
µg/dL
  Baseline (Week 8) to Week 16 | 33.77 [-160.13 to 229.67] | 245.50 [-102.60 to 593.60]
  Week 16 to Week 20 | -7.30 [-253.61 to 239.02] | -244.20 [-711.30 to 222.80]
  Week 20 to Week 24 | 53.40 [-239.71 to 346.51] | 88.80 [-429.40 to 606.90]

4. Secondary Outcome: Change Over Time in Threat Bias Score From Dot Probe Task
Description: Changes in threat bias scores assessed using Dot Probe task during labs at weeks 8, 16, 20 and 24. The bias measurement protocol consists of 144 trials (48 threat congruent, 48 threat incongruent, 48 neutral presentations). Participants indicate the probe letter via button press. Angry face location, probe location, probe type and actor are all fully counterbalanced in presentation. The threat bias score equals the mean of reaction time on threat congruent from threat incongruent trials. A threat bias scores >0 indicate a bias towards threat, whereas scores <0 mean that the participant is slower to respond to threatening stimuli than neutral stimuli. Reaction times were measured in milliseconds. Change over time is defined as the difference in least square means between timepoints with 95% confidence interval limits.
Time Frame: up to 24 weeks
Population: Data reported from tasks completed.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliseconds
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Number analyzed (Participants) | 34 | 41
milliseconds
  Baseline (Week 8) to Week 16 | -5.23 [-21.51 to 11.06] | -3.75 [-14.95 to 7.45]
  Week 16 to Week 20 | -2.49 [-19.75 to 14.78] | -3.81 [-15.79 to 8.16]
  Week 20 to Week 24 | -0.92 [-18.31 to 16.47] | 7.25 [-4.67 to 19.17]

5. Secondary Outcome: Change Over Time in Percent of "Hard Task" Choice in EEfRT
Description: Effort Expenditure for Rewards Task (EEfRT) measures approach motivation that indexes the willingness to expend effort to obtain monetary rewards under varying conditions of reward probability and magnitude. On each trial, participants choose between an "easy task" and a "hard task" and are presented with information about the probability of winning (i.e., 12%, 50%, or 88%), and the magnitude of the potential reward if they complete the button-press task successfully (range: $1.24 - $4.12). Completion of the easy task requires 30 button presses in 7 seconds using the dominant index finger, whereas completion of the hard task requires 100 presses with the non-dominant "pinky" finger in 21 seconds. The percent of hard task choices is the dependent measure. Change over time is defined as the difference in least square means between time points with 95% confidence interval limits.
Time Frame: up to 24 weeks
Population: Data reported from tasks completed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of "hard task" choices
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
Number analyzed (Participants) | 38 | 36
percentage of "hard task" choices
  Baseline (Week 8) to Week 16 | -0.0044 [-0.1306 to 0.1219] | 0.0086 [-0.0870 to 0.1042]
  Week 16 to Week 20 | 0.0019 [-0.1309 to 0.1347] | 0.0289 [-0.0720 to 0.1298]
  Week 20 to Week 24 | -0.0045 [-0.1392 to 0.1303] | 0.0200 [-0.0885 to 0.1286]

ADVERSE EVENTS:
Time Frame: From Baseline (Week 8) through study Week 24, an approximate total of 16 weeks.
Arm/Group | Placebo Patch and Placebo Capsule | Estradiol Patch and Progesterone Capsule
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 39/40 | 39/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Patch and Placebo Capsule (N=40) | Estradiol Patch and Progesterone Capsule (N=42)
Breast tenderness (Reproductive system and breast disorders) | 11 (16) | 30 (91)
Profuse menstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 10 (13) — Profuse is defined as >3 tampons or pads for > 5 days or > 1 tampon or pad per hour on any given day.
Prolonged menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 5 (5) — Menstrual bleeding > 10 days.
Headache (Non-Migraine) (Nervous system disorders) | 29 (75) | 27 (63)
Migraine (Nervous system disorders) | 5 (8) | 3 (4)
Negative Mood Change (Psychiatric disorders) | 17 (37) | 17 (27)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 (29) | 12 (20)
Nausea (Gastrointestinal disorders) | 12 (14) | 15 (24)
Skin irritation (at patch site) (Skin and subcutaneous tissue disorders) | 18 (36) | 33 (96)
Hypertension (Cardiac disorders) | 3 (4) | 8 (10)
Weight gain (Metabolism and nutrition disorders) | 4 (7) | 0 (0)
Lightheadedness (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03003949/Prot_SAP_000.pdf